CLINICAL TRIAL: NCT01143714
Title: A Vehicle-Controlled Study to Determine the Effect of Four Weeks of Debridement With Collagenase Santyl Ointment (Santyl) on the Healing of Diabetic Foot Ulcers
Brief Title: A Study to Look at the Effects of Four Weeks of Treatment on the Healing of Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 017-101-09-024
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Collagenases; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Santyl
- B (Placebo Comparator)
  Interventions: Other: White Petrolatum

INTERVENTIONS:
Drug: Santyl — Apply an amount sufficient (thickness of a nickel) to cover the wound area. It will be applied once daily during the treatment phase, up to four weeks.
  Arms: A
Other: White Petrolatum — Apply an amount sufficient (thickness of a nickel) to cover the wound area. It will be applied once daily during the treatment phase, up to four weeks.
  Arms: B

SUMMARY:
The purpose of this study is to assess the effect of four weeks of treatment with Santyl Ointment, compared to White Petrolatum, on the change from baseline in wound area of diabetic foot ulcers over four weeks, and on the proportion of subjects achieving complete wound closure within 12 weeks from initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent document Photography Release must be read, signed, and dated by the subject or the subject's legally authorized representative before conducting any study procedures or exams. In addition, the informed consent document must be signed and dated by the individual who consents the subject before conducting the screening visit. A photocopy of the signed informed consent document must be provided to the subject, and the original signed document placed in the subject's chart.
* Age 18 years and older. Subjects may be of either sex and of any race or skin type.
* Women of child-bearing potential (those who are not premenarchal, not surgically sterilized [hysterectomy or bilateral oophorectomy], or not post-menopausal) may participate in the study if they meet all of the following conditions:

  * they are not breast feeding
  * undertake an HCG serum pregnancy test, which must be negative
  * they do not intend to become pregnant during the study
  * they are using adequate birth control methods and they agree to continue using those methods for the duration of the study
* Post-menopausal is defined as no period in the previous 12 months Adequate birth control methods are defined as: hormonal-topical, oral, implantable or injectable contraceptives; mechanical-spermicide in conjunction with a barrier such as a condom or diaphragm; IUD; or, surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use an adequate birth control method as described above for the remainder of the study.

NOTE: Women who have had a bilateral tubal ligation are not considered to have been surgically sterilized and must agree to the conditions as specified above.

* Willing to make all required study visits and to use the Darco shoe off-loading device and insole.
* Able to follow instructions, particularly regarding the application of test articles and dressings at home. Able to apply the test article, or has a caregiver available to apply the test article according to the protocol.
* Have a diabetic foot ulcer, Wagner Grades† 1 or 2, on the plantar surface of the foot.
* Target ulcer present for at least 28 days, but no longer than 18 months, and has failed to close by ≥ 40% during the first 4 weeks of therapy administered during the past 4 to 8 weeks.
* Target ulcer area between 2 and 15 cm², post debridement, if required. 9- Adequate arterial blood flow as evidenced by an ankle brachial index (ABI) of > 0.7 and ≤ 1.1; if the ABI is greater than 1.1, then a toe pressure of > 30 mmHg OR a TcPO2 ≥ 40 mmHg; either secondary measure is acceptable, but if both are obtained, each must meet its respective cutoff.
* 10. Reasonable control of blood glucose, as evidenced by a serum HbA1C ≤ 12% at screening.
* 11.Acceptable state of health and nutrition as evidenced by a serum pre-albumin level ≥ 15 mg/dL (0.15 g/L) and serum albumin ≥ 2.0 g/dL (20 g/L) at screening.
* 12. Hematology values in the following ranges: WBC ≥ 3.0x109/L Hgb ≥ 10.0 g/dL Neutrophils ≥ 1.5x109/L Platelets ≥ 75 x109/L Normal blood smear
* Blood chemistry values and urinalysis in the following ranges (Healthpoint Ranges):

Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) Alkaline phosphatase ≤ 2.5 times the ULN Alanine transaminase (ALT) ≤ 2.5 times the ULN Aspartate transaminase (AST) ≤ 2.5 times the ULN Serum creatinine ≤ 1.5 times the ULN Urinalysis: WBC < 4/HPF; RBC < 4/HPF

Exclusion Criteria:

* Contraindications or known hypersensitivity to the test articles or their components.
* Therapy with another investigational agent within 30 days, lower extremity angioplasty within 4 weeks, untreated osteomyelitis, or chemotherapy or radiation therapy within 5 years prior to screening.
* Prior therapy of the target wound with Santyl.
* Current therapy with systemic antibiotics to treat a foot ulcer, or prescription topical antibiotics on the target ulcer.
* Target ulcer located over the heel (talus, distal calcaneous, navicular, or cuboid).
* Fracture of bones in the target ulcer foot occurring within the past 3 months.
* Cellulitis or abscess of the target ulcer foot.
* A positive result from the screening Quantitative Bacteriology (Qbac) biopsy. A wound will be considered infected if the laboratory findings reveal ≥ 106 colony forming units (cfu) per gram of tissue or > 1 beta-hemolytic Streptococcus per gram of tissue.
* Target ulcer tunneling, per probing.
* More than three DFU on the target foot. The target ulcer must be at least 2 cm from another ulcer.
* Concomitant severe burn, immunodeficiency disorder, hematologic disorder, or malignancy (other than non-melanoma skin cancer) beyond the in situ stage.
* Abnormal laboratory values that, in the opinion of the Principal Investigator, place the subject at risk for the study.
* Positive serum HCG pregnancy test.
* The Medical Monitor may declare any subject ineligible for a valid procedural or medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint
Locations (6):
- United States (6):
  - Olive View - UCLA Medical Center, Sylmar, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - The Foot and Ankle Institute of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Center for Advanced Wound Care, Wyomissing, Pennsylvania
  - Complete Family Foot Care, McAllen, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults aged 18 years and older, with a diabetic foot ulcer that has not responded to treatment
Groups:
- Collagenase Santyl Ointment: Santyl : Applied an amount sufficient (thickness of a nickel) to cover the wound area. It will be applied once daily during the treatment phase, up to four weeks.
- Vehicle (White Petrolatum): White Petrolatum : Applied an amount sufficient (thickness of a nickel) to cover the wound area. It will be applied once daily during the treatment phase, up to four weeks.
Period: Overall Study
Arm/Group | Collagenase Santyl Ointment | Vehicle (White Petrolatum)
Started | 29 | 28
Completed | 22 | 25
Not Completed | 7 | 3
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Subject non-compliance | 0 | 1
Not completed — wound closed = deemed healed | 1 | 0
Not completed — wound size increased | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Collagenase Santyl Ointment | Vehicle (White Petrolatum) | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 9 | 9 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.4) | 59.9 (12.4) | 59.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 21 | 23 | 44
Region of Enrollment [Number; unit: participants]
  United States | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change in Wound Area
Description: The primary efficacy endpoint was the percent change in wound area from baseline to completion of the 4-week treatment phase and the 8-week follow-up period
Time Frame: 4 Weeks
Population: Sample size originally set at 100 to provide 80% power, a=0.05. Interim analysis when enrollment reached 50 indicated results would not change with additional enrollment. Intent-to-treat used for primary inference; Missing values imputed by method of population mean and last observation carried forward (wound area).
Measure: Least Squares Mean (Standard Error); unit: percentage of average change in wound
Arm/Group | Collagenase Santyl Ointment | Vehicle (White Petrolatum)
Number analyzed (Participants) | 29 | 28
percentage of average change in wound
  Treatment Phase | -32.74 (7.12) | -33.08 (7.13)
  Follow-up Period | -49.34 (12.34) | -34.27 (12.36)

2. Secondary Outcome: Number of Sharp Debridements Performed During the 4-week Treatment Phase and the 8-week Follow-up Period (12 Weeks Total)
Time Frame: 12 weeks
Population: Intent-to-Treat population
Measure: Least Squares Mean (Standard Error); unit: debridements
Arm/Group | Collagenase Santyl Ointment | Vehicle (White Petrolatum)
Number analyzed (Participants) | 29 | 28
debridements | 1.38 (0.22) | 1.5 (0.22)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Covered both 4 week treatment phase and the 8 week follow-up period.
Arm/Group | Collagenase Santyl Ointment | Vehicle (White Petrolatum)
Serious Adverse Events (participants affected / at risk) | 4/29 | 4/28
Other Adverse Events (participants affected / at risk) | 1/29 | 5/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collagenase Santyl Ointment (N=29) | Vehicle (White Petrolatum) (N=28)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Necrotizing Fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collagenase Santyl Ointment (N=29) | Vehicle (White Petrolatum) (N=28)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release.